CLINICAL TRIAL: NCT05762328
Title: Adherence to Clinical Guidelines Regarding the Duration of Antibiotic Treatment in Patients Hospitalized for Community-acquired Pneumonia With Clinical sTability. ADAPT Study
Brief Title: Duration of Antibiotic Treatment in Community-acquired Pneumonia
Acronym: ADAPT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto de Investigacion Sanitaria La Fe (Other)
Collaborators: Instituto de Salud Carlos III (Other Government); Sociedad Española de Neumología y Cirugía Torácica (Other); Sociedad Valenciana de Neumología (Unknown)
Responsible Party: Principal Investigator, Raúl Méndez, MD PhD, Dr., Instituto de Investigacion Sanitaria La Fe
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2022-914-1
Record Dates: First submitted 2023-02-28; First posted 2023-03-09 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2024-01

CONDITIONS: Community-acquired Pneumonia
Keywords: pneumonia; antibiotic treatment; duration; clinical stability; adherence
MeSH Terms: conditions — Community-Acquired Pneumonia; Pneumonia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of care (No Intervention): Patients allocated in hospitals randomized to non-interventional arm. Observational analysis of patients treated by clinicians with standard of care.
- Interventional (Other): Patients allocated in hospitals randomized to interventional arm. Intervention: automatic reminders through pop-up windows in the computerized prescription software, reminding the clinician responsible for each patient of the need to adhere to clinical guidelines regarding the duration of antibiotic treatment in patients with clinical stability
  Interventions: Behavioral: Reminders to the assistant clinicians of the need to adhere to clinical guidelines regarding the duration of antibiotic treatment community-acquired pneumonia

INTERVENTIONS:
Behavioral: Reminders to the assistant clinicians of the need to adhere to clinical guidelines regarding the duration of antibiotic treatment community-acquired pneumonia — Automatic reminders through pop-up windows in the computerized prescription software, reminding the clinician responsible for each patient of the need to adhere to clinical guidelines regarding the duration of antibiotic treatment in patients with clinical stability
  Other Names: Reminders to the clinician responsible for each patient of the need to adhere to clinical guidelines regarding the duration of antibiotic treatment in patients with clinical stability
  Arms: Interventional

SUMMARY:
International and national clinical guidelines recommend short antibiotic regimens in patients with non-severe community-acquired pneumonia (CAP) who have reached clinical stability. However, adherence to these recommendations remains unclear. The goals of this quasi-experimental trial are: 1) to assess adherence to clinical guidelines in relation to the duration of antibiotic treatment in patients hospitalized for non-severe CAP who have reached clinical stability; 2) increase adherence to clinical guidelines and reduce the use of antibiotics in patients hospitalized for non-severe CAP who have achieved clinical stability after at least 5 days of antibiotic treatment.

To this end, a multicenter prospective study will be carried out over 2 years and divided into 2 phases: i) during the first year (observational phase), patients with CAP hospitalized in the participating centers will be recorded to assess objective 1; ii) to achieve objective 2, at the beginning of the second year (quasi-experimental trial) the centers will be randomized into 2 groups of hospitals, one of them a control group and the other an intervention group. The intervention will consist in automatic reminders through pop-up windows in the computerized prescription software, reminding the clinician responsible for each patient of the need to adhere to clinical guidelines regarding the duration of antibiotic treatment in patients with clinical stability.

ELIGIBILITY:
Inclusion Criteria:

* Patients >18 years hospitalized for community-acquired pneumonia with a new infiltrate on chest X-ray and/or computerized tomography.
* At least one compatible sign or symptom (fever, cough, expectoration, dyspnea, chest pain or crackles on auscultation)
* Correctly treated with ≥ 3 days of antibiotic

Exclusion Criteria:

* Intensive care unit admission during the first 5 days since hospital admission
* Abscess or necrotizing pneumonia
* Empyema or pleural effusion requiring drainage tube
* Bronchiectasis
* Cystic fibrosis
* Active tuberculosis
* Postobstructive pneumonia
* Suspected bronchial aspiration
* SARS-CoV-2 infection
* Immunosuppression (congenital immunodeficiencies, HIV infection, solid organ transplantation, functional or anatomical asplenia, immunosuppressive treatment, active solid or haematological neoplasia [active treatment in the last 12 months], etc.)
* Hospital acquired pneumonia
* Concomitant extrapulmonary infection that requires antibiotic treatment for more than 5 days (eg myocarditis)
* Confirmed diagnosis alternative to pneumonia (eg, lung cancer)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Duration of antibiotic treatment | 90 days
  Total duration in days of antibiotic treatment (including the days of outpatient antibiotic prescribed at discharge).

SECONDARY OUTCOMES:
Duration of antibiotic treatment after reaching clinical stability | 90 days
  Duration in days of antibiotic treatment after reaching clinical stability
Patients treated with an adequate duration of 5±1 days | 90 days
  Percentage of patients treated with an adequate duration of 5±1 days
Patients admitted to the ICU after the 5th day | 90 days
  Percentage of patients admitted to the ICU after the 5th day of admission
Mortality | 90 days
  Percentage of patients who died during the study
Readmission | 90 days
  Percentage of patients who are readmitted after hospital discharge
Reintroduction of antibiotic treatment | 90 days
  Percentage of patients with reintroduction of antibiotic treatment
Length of hospital stay | 90 days
  Length of hospital stay in days
Adverse events related to antibiotic treatment | 90 days
  Percentage of patients with adverse events related to antibiotic treatment

OTHER OUTCOMES:
Factors related to excess of antibiotic treatment | 90 days
  Factors o variables related to excess of antibiotic treatment

CONTACTS AND LOCATIONS:
Overall Officials: Raúl Méndez, MD, PhD, Principal Investigator — Instituto de Investigación Sanitaria La Fe
Locations (1):
- University and Polytechnic Hospital La Fe, Valencia, Spain

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, CSR